CLINICAL TRIAL: NCT01869569
Title: Effect of Pregabalin in Patients With Radiotherapy-Related Neuropathic Pain: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Pregabalin in Patients With Radiotherapy-related Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012026; SYSN002 (Other: Sun Yat-sen Memorial Hospital, Neurology department)
Record Dates: First submitted 2013-05-26; First posted 2013-06-05 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Neuropathic Pain
Keywords: Radiation; Neuropathic Pain; Pregabalin
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Active Comparator): Arm I:At the 4-week dose-titration phase, will receive one capsule of pregabalin (75 mg) twice daily from Day 1 to Day 7, and two capsules of pregabalin (150 mg) twice daily from Day 8 to Day 14. From Day 15 to Day 28, patients will perform dosage adjustments based on the pain relief and tolerability. At maintenance phase, patients will take the optimized dosage of pregabalin.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Arm II:At the 4-week dose-titration phase, will receive one capsule of placebo twice daily from Day 1 to Day 7, and two capsules of placebo twice daily from Day 8 to Day 14. From Day 15 to Day 28, patients will perform dosage adjustments based on the pain relief and tolerability. At maintenance phase, patients will take the optimized dosage of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — At the 4-week dose-titration phase, will receive one capsule of pregabalin (75 mg) twice daily from Day 1 to Day 7, and two capsules of pregabalin (150 mg) twice daily from Day 8 to Day 14. From Day 15 to Day 28, patients will perform dosage adjustments based on the pain relief and tolerability. At maintenance phase, patients will take the optimized dosage of pregabalin.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — At the 4-week dose-titration phase, will receive one capsule of placebo twice daily from Day 1 to Day 7, and two capsules of placebo twice daily from Day 8 to Day 14. From Day 15 to Day 28, patients will perform dosage adjustments based on the pain relief and tolerability. At maintenance phase, patients will take the optimized dosage of placebo.
  Arms: Placebo

SUMMARY:
Rationale: Pregabalin is effective on radiotherapy-related neuropathic pain. Purpose: This randomized, double-blind, placebo-controlled trial aims to investigate the effect and safety of pregabalin in treating radiotherapy-related neuropathic pain.

DETAILED DESCRIPTION:
Radiotherapy for cancer is associated with peripheral neuropathies, especially with brachial plexus neuropathy and trigeminal neuralgia, which included painful sensation that are described as burning, aching, spasm, or tingling. Though there is some recommendation about neuropathic pain, there is no definite drug which is recommended for radiotherapy-related neuropathic pain.

Pregabalin, a central nervous system(CNS)-active compound, is an analog of the neurotransmitter gamma-aminobutyric acid. It has been proved an effective treatment for diabetic peripheral neuropathy and postherpetic neuralgia in previous clinical trials. This study plans to evaluate the efficacy of pregabalin versus placebo for relieving radiotherapy-related peripheral neuropathic pain, and assessed its safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received radiation therapy for histologically confirmed head and neck cancer.
2. Clinical evidence support the diagnosis of radiation-related neuropathic pain (confirmed by the Michigan Neuropathy Screening Instrument) and had a daily pain score of 4 or higher based on a numerical rating scale (0-10 points).
3. Neuropathic pain defined according to clinical history, symptoms, physical signs, and a score>= 12 in Chinese version of Leeds Assessment of Neuropathic Symptoms and Signs questionnaire by two neurology specialists.
4. The mean duration of pain is more than 4 weeks.
5. Fertile women who are willing to take contraception during the trial.
6. Routine laboratory studies with bilirubin </=2 * upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) < 2 * ULN, creatinine <1.0 * ULN, red-cell count >/= 4,000 per cubic millimeter; white-cell count >/=1500 per cubic millimeter, platelets >/= 75,000 per cubic millimeter; Hb >/=9.0.
7. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Current diagnosis of tumor recurrence or metastasis and evidence of tumor associated pain.
2. Evidence of secondary neuropathic pain other than radiation.
3. Treatment with carbamazepine, gabapentin or pregabalin within 30 days before study enrollment.
4. Ongoing treatment for neuropathic pain.
5. History of anaphylactic response to pregabalin.
6. Evidence of sever systematic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) at week 16 | week 16
  The primary efficacy measure is the reduction of NRS from baseline to week 16.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | week 16
  The investigators compare the BPI scores at week 16 with those at baseline.
the Profile of Mood States-Short Form (POMS-SF) | week 16
  The investigators compare the POMS-SF scores at week 16 with those at baseline.
the World Health Organization Quality of Life-BREF (WHOQOL-BREF) | week 16
  The investigators compare the WHOQOL-BREF scores at week 16 with those at baseline.
Patient Global Impression of Change (PGIC) | week 16
  Number of Participants With Treatment Success at the End of Therapy as Measured by the Patient Global Impression of Change (PGIC). A treatment success is defined as Much or Very Much Improved at the Week 16. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improved
Clinical Global Impression of Change (CGIC) | week 16
  Number of Participants With Treatment Success at the End of Therapy Based on Clinical Global Impression of Change (CGIC) . A treatment success is defined as Much or Very Much Improved at the Week 16. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improve.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D.,PhD., Principal Investigator — Department of Neurology, Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Huiai Hospital, Guangzhou, Guangdong
  - Zengcheng People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang J, Li Y, Shen Q, Rong X, Huang X, Li H, Zhou L, Mai HQ, Zheng D, Chen MY, Xu Y, Li J, Hui X, Simone CB 2nd, Gaertner J, Argyriou AA, Chow E, Chen P, Tang Y. Effect of Pregabalin on Radiotherapy-Related Neuropathic Pain in Patients With Head and Neck Cancer: A Randomized Controlled Trial. J Clin Oncol. 2019 Jan 10;37(2):135-143. doi: 10.1200/JCO.18.00896. Epub 2018 Nov 20. PMID 30457920